CLINICAL TRIAL: NCT00001978
Title: Determination of Glomerular Filtration Rate, Effective Renal Plasma Flow and Glomerular Capillary Wall Permselectivity
Brief Title: Determination of Kidney Function
Status: Terminated | Type: Observational
Why Stopped: All analysis with identifiable specimens/data is complete or site has no identifiers linked to the specimens/data
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 890152; 89-DK-0152
Record Dates: First submitted 2000-01-20; First posted 2000-01-21 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Kidney Disease; Proteinuria; Autoimmune / Connective Tissue Diseases
Keywords: Kidney Disease; Kidney Function Tests; Proteinuria
MeSH Terms: conditions — Kidney Diseases; Proteinuria; Connective Tissue Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Study Cohort: Selected patients with proteinuria

SUMMARY:
Much more about kidney disorders can be learned by determining kidney function. This research proposes to study the kidneys function by several parameters known as glomerular filtration rate (GFR), Renal Plasma Flow (RPF), and Glomerular Capillary Wall Permselectivity.

The study will select patients suffering from different types of kidney diseases. These patients will be selected based on the presence of significant amounts of protein in their urine (proteinuria).

Standard blood and urine tests are often unable to provide completely accurate information about the kidney. In order for researchers to have a more accurate idea of kidney function, they will use alternative tests. Test materials (para aminohippurate and inulin) will be injected into patients veins that provides information based on their filtration through the kidneys....

DETAILED DESCRIPTION:
The study of various kidney disorders will be facilitated by determinations of true glomerular filtration rate and/or effective renal plasma flow employing inulin or non-radioactive iothalamate and/or para aminohippurate (PAH), respectively.

Selected patients with proteinuria will be asked to participate in studies of glomerular capillary wall permselectivity calculated from the fractional clearances of the endogenous proteins, albumin and IgG and from the fractional clearances of polydisperse neutral dextran with effective molecular radii ranging from 20-60 angstroms. To achieve this, low molecular weight dextran will be administered by slow IV injection immediately following the inulin or iothalamate and/or PAH priming doses.

Glomerular filtration rate, effective renal plasma flow and/or glomerular permselectivity can be measured simultaneously during a standard hydrated urinary clearance study. Timed urine and blood collections will be obtained, typically requiring a total of 60 to 90 minutes. The total test time, including pre-test hydration, is 4 to 5 hours.

Alternatively, glomerular filtration rate can be measured by one of two plasma clearance methods that do not require urine collections. For one method, a steady-state plasma concentration of iothalamate will be achieved in ambulatory patients by a 24-hour subcutaneous infusion of iothalamate using an insulin pump. For the second method, the decline in plasma concentration of iothalamate will be measured after an intravenous dose of iothalamate.

ELIGIBILITY:
* INCLUSION CRITERIA:

Ability to provide informed assent to all aspects of the study after full information is provided.

An indication to measure kidney function as accurately as possible in the context of an approved clinical protocol within the intramural programs of the National Institutes of Health:

* For minor subjects, a clinical indication will be required.
* For adult subjects, a clinical and/or research indication will be required.

EXCLUSION CRITERIA:

Pregnant females or nursing mothers will be excluded from all aspects of this study (at least until the infant is stable on a regimen of formula feeding).

Patients will not receive a test material if there is a history of allergy to that material.

Patients with a history of bronchial asthma or allergy to iodine-containing contrast material will not receive iothalamate.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary clinical and community sample
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 1989-10-11 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate | 4-5 hours
  Glomerular filtration rate, effective renal plasma flow and /or glomerular permselectivity can be measured simultaneously during astandard hydrated urinary clearance study. Timed urine and blood collections will be obtained, typically requiring a total of 60 to 90 minutes. The total test time, including pretest hydration, is 4 to 5 hours.

SECONDARY OUTCOMES:
Effective renal plasma flow
  Glomerular filtration rate, effective renal plasma flow and /or glomerular permselectivity can be measured simultaneously during astandard hydrated urinary clearance study. Timed urine and blood collections will be obtained, typically requiring a total of 60 to 90 minutes. The total test time, including pretest hydration, is 4 to 5 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Meryl A Waldman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Shemesh O, Golbetz H, Kriss JP, Myers BD. Limitations of creatinine as a filtration marker in glomerulopathic patients. Kidney Int. 1985 Nov;28(5):830-8. doi: 10.1038/ki.1985.205. PMID 2418254
- [Background] Bauer JH, Brooks CS, Burch RN. Clinical appraisal of creatinine clearance as a measurement of glomerular filtration rate. Am J Kidney Dis. 1982 Nov;2(3):337-46. doi: 10.1016/s0272-6386(82)80091-7. PMID 7148824
- [Background] Blythe WB. The endogenous creatinine clearance. Am J Kidney Dis. 1982 Nov;2(3):321-3. doi: 10.1016/s0272-6386(82)80089-9. No abstract available. PMID 7148823
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1989-DK-0152.html